CLINICAL TRIAL: NCT02506842
Title: A Prospective, Multi-centric, Phase Ⅲ, Randomized, Controlled Study to Evaluate the Efficacy and Safety of Second-Line Adjuvant Therapy With Nab-Paclitaxel Plus Gemcitabine (AG) Versus Oxaliplatin Plus Folinic Acid and Fluorouracil (OFF) for Gemcitabine-Refractory Pancreatic Cancer After Curative Resection
Brief Title: Second-Line Adjuvant Therapy With Nab-Paclitaxel Plus Gemcitabine Versus Oxaliplatin Plus Folinic Acid and Fluorouracil for Gemcitabine-Refractory Pancreatic Cancer After Curative Resection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, M.D PH.D, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPAC-010
Record Dates: First submitted 2015-07-18; First posted 2015-07-23 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Stage ⅠA Pancreatic Cancer; Stage ⅠB Pancreatic Cancer; Stage ⅡA Pancreatic Cancer; Stage ⅡB Pancreatic Cancer
Keywords: Pancreatic Cancer; Pancreatic Adenocarcinoma; AG; OFF; Second-Line Adjuvant Therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nab-paclitaxel + gemcitabine (AG) (Experimental): nab-paclitaxel at 100 mg/m^2 on days 1, 8, and 15; gemcitabine at 1000 mg/m^2 on days 1, 8, and 15
  Interventions: Drug: nab-paclitaxel; Drug: gemcitabine
- oxaliplatin + folinic acid + fluorouracil (OFF) (Experimental): oxaliplatin at 85mg/m^2 on days 8 and 22, folinic acid at 200mg/m^2 on days 1,8,15 and 22, fluorouracil at 2000mg/m^2 on days 1,8,15 and 22.
  Interventions: Drug: oxaliplatin; Drug: folinic acid; Drug: fluorouracil

INTERVENTIONS:
Drug: nab-paclitaxel — Patients firstly receive nab-paclitaxel 100 mg/m^2 (iv, 30 minutes) on days 1, 8, and 15 for 3 weeks, followed by one week without treatment. Treatment repeats until there is disease progression or recurrence.
  Other Names: Abraxane
  Arms: nab-paclitaxel + gemcitabine (AG)
Drug: gemcitabine — Patients secondly receive gemcitabine 1000 mg/m^2 (iv, 30 minutes) on days 1, 8, and 15 for 3 weeks, followed by one week without treatment. Treatment repeats until there is disease progression or recurrence.
  Other Names: GEMZAR
  Arms: nab-paclitaxel + gemcitabine (AG)
Drug: oxaliplatin — Patients receive oxaliplatin 85 mg/m^2 (iv, 2 hours) on days 8 and 22 with 42 days as a cycle. Treatment repeats until there is disease progression or recurrence. Oxaliplatin is given before folinic acid and fluorouracil when the three drugs are given on the same days.
  Arms: oxaliplatin + folinic acid + fluorouracil (OFF)
Drug: folinic acid — Patients receive folinic acid 200 mg/m^2 (iv) on days 1, 8, 15 and 22 for 4 weeks, followed by 2 weeks without treatment. Treatment repeats until there is disease progression or recurrence.
  Other Names: LV
  Arms: oxaliplatin + folinic acid + fluorouracil (OFF)
Drug: fluorouracil — Patients receive fluorouracil 2000 mg/m^2 (iv, 24 hours) on days 1, 8, 15 and 22 for 4 weeks, followed by 2 weeks without treatment. Treatment repeats until there is disease progression or recurrence.
  Arms: oxaliplatin + folinic acid + fluorouracil (OFF)

SUMMARY:
The purpose of this study is to investigate the activity and safety of second-line adjuvant therapy with nab-paclitaxel plus gemcitabine (AG) versus oxaliplatin plus folinic acid and fluorouracil (OFF) for gemcitabine-refractory pancreatic cancer after curative resection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* To evaluate the therapeutic efficacy of second-line adjuvant therapy with nab-paclitaxel plus gemcitabine (AG) versus oxaliplatin plus folinic acid and fluorouracil (OFF) in terms of overall survival for gemcitabine-refractory pancreatic cancer after curative resection.

SECONDARY OBJECTIVES:

* To evaluate the therapeutic efficacy of two regimens in terms of objective response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* To evaluate the time to remission of patients treated with the two regimens.
* To evaluate the progression-free survival of patients treated with the two regimens.
* To evaluate the levels of tumor biomarkers in serum of patients treated with the two regimens, including Carbohydrate Antigen (CA)19-9、CA125、CA153、CA242、CA72-4、CA50、CEA、AFP.
* To evaluate the occurrence of grade 3 and 4 toxicities according to National Cancer Institute Common Toxicity Criteria for Adverse Effects (NCI CTCAE) version 4.0 in patients treated with the two regimens.
* To evaluate the quality of life score of patients treated with the two regimens.

Detailed Description of Arms:

Patients are randomized to 1 of 2 treatment arms (Arm AG or Arm OFF). Arm AG: Firstly, patients receive nab-paclitaxel 100 mg/m^2 (iv, 30 minutes) on days 1, 8, and 15 for 3 weeks, followed by one week without treatment. Secondly, patients receive gemcitabine 1000 mg/m^2 (iv, 30 minutes) on days 1, 8, and 15 for 3 weeks, followed by one week without treatment. Treatment repeats until there is disease progression or recurrence.

Arm OFF: Patients receive oxaliplatin 85 mg/m^2 (iv, 2 hours) on days 8 and 22 with 42 days as a cycle. Patients receive folinic acid 200 mg/m^2 (iv) and fluorouracil 2000 mg/m^2 (iv, 24 hours) on days 1, 8, 15 and 22 for 4 weeks, followed by 2 weeks without treatment. Oxaliplatin is given before folinic acid and fluorouracil when the three drugs are given on the same days. Treatment repeats until there is disease progression or recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed content obtained prior to treatment
* Age ≥ 18 years and ≤ 75 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must have histologically confirmed pancreatic adenocarcinoma (or any mixed pathology if adenocarcinoma is predominant) after R0 or R1 resection. The pathological staging does not exceed the stage ⅡB. And the patients have received gemcitabine as adjuvant chemotherapy after curative resection.
* There is progression or recurrence of tumor during the course of adjuvant chemotherapy with gemcitabine, or within 6 months after the whole courses of treatment.
* No severe defects in hematological system, immune system, cardiac function and pulmonary function.
* White blood cell (WBC) ≥ 4 × 10^9/L; Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L; Platelets (PLT) ≥ 100 × 10^9/L; Hemoglobin (Hgb) ≥ 9 g/dL
* Aspartate aminotransferase (AST) (serum glutamate oxaloacetate transaminase (SGOT)）/ alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase (SGPT)) ≤ 2.5 × institutional upper limit of normal (ULN); Total bilirubin (TBIL) ≤ ULN; Creatinine (CRE) ≤ 1.5 × ULN
* Prothrombin time (PT) and international normalized ratio (INR) ≤ 1.5 × ULN
* The patients are willing to comply to the study plan and other requirements.

Exclusion Criteria:

* There is another malignant tumor with the patient.
* Patients who have received any form of anti-tumor therapy within 4 weeks prior to the enrollment, including chemotherapy, radiotherapy, interventional chemoembolization, radiofrequency ablation, and molecular targeted therapy
* Use of any other investigational agents within 4 weeks prior to the enrollment.
* The progression or recurrence of tumor occurs after 6 months of the course of the adjuvant chemotherapy with gemcitabine.
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, internal hemorrhage, pancreatic leakage, bile leakage, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of allergic reactions attributed to compounds of similar chemical or biological composition to the drugs.
* Metabolic acidosis, acute or chronic, including ketoacidosis
* Pregnant or nursing women
* Any event or condition that is possible to harm the safety of the patients or the integrities of data, including severe medical risk factors, medical conditions, and laboratory disorders.
* Patients who are unwilling or unable to comply with study procedures, or may be absent from the observation for more than 7 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of enrollment until the date of death from any cause, assessed 2 cycles during the therapy and 3 months thereafter up to 24 months; Cycle 1 (each cycle is 28 days for AG regimen and 42 days for OFF regimen).
  To evaluate the therapeutic efficacy of second-line adjuvant therapy with AG versus OFF in terms of overall survival for gemcitabine-refractory pancreatic cancer after curative resection. Outpatient visit, phone interview

SECONDARY OUTCOMES:
Objective Response Rate | Complete Remission% + Partial Remission %, assessed 2 cycles during the therapy and 3 months thereafter up to 24 months; Cycle 1 (each cycle is 28 days for AG regimen and 42 days for OFF regimen).
  To evaluate the therapeutic efficacy of two regimens in terms of objective response rate. Computed tomography (CT) scan
Time to Remission | From date of enrollment until the date of remission, assessed 2 cycles during the therapy and 3 months thereafter up to 24 months; Cycle 1 (each cycle is 28 days for AG regimen and 42 days for OFF regimen).
  To evaluate the time to remission of patients treated with the two regimens. Computed tomography (CT) scan
Progression-Free Survival | From date of enrollment until the date of first documented progression, assessed 2 cycles during the therapy and 3 months thereafter up to 24 months; Cycle 1 (each cycle is 28 days for AG regimen and 42 days for OFF regimen).
  To evaluate the progression-free survival of patients treated with the two regimens. Computed tomography (CT) scan
The Levels of Tumor Biomarkers in Serum | 2 cycles during the therapy and 3 months thereafter up to 24 months; Cycle 1 (each cycle is 28 days for AG regimen and 42 days for OFF regimen).
  To evaluate the levels of tumor biomarkers in serum of patients treated with the two regimens, including Carbohydrate Antigen (CA)19-9、CA125、CA153、CA242、CA72-4、CA50、CEA、AFP . Outpatient visit, laboratory findings
Number of grade 3 and 4 toxicities according to NCI CTCAE version 4.0 | 1 week during therapy and 3 months thereafter up to 24 months.
  To evaluate the occurrence of grade 3 and 4 toxicities according to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE; version 4.0) in patients treated with the two regimens. The toxicity profile includes but not limits neutropenia, thrombocytopenia, peripheral neuropathy, hypoglycemia, metabolic acidosis (acute or chronic, including ketoacidosis), which will be summarized as the percentage of patients by type and grade according to treatment group. Outpatient visit, laboratory findings.
Quality of life | 2 cycles during the therapy and 3 months thereafter up to 24 months; Cycle 1 (each cycle is 28 days for AG regimen and 42 days for OFF regimen).
  To evaluate the quality of life score of patients treated with the two regimens. Outpatient visit, phone interview

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Jun Yu, M.D PH.D, Principal Investigator — Department of Pancreatic and Hepatobiliary Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University; 270 Dong An Road, Shanghai 200032, China
Locations (7):
- China (7):
  - Department of Hepatobiliary Surgery, Sun Yat-Sen University Cancer Center,Sun Yat-Sen University, Guangzhou, Guangdong
  - Department of Biliary Pancreatic Surgery, Shanghai Changzheng Hospital, The Second Military Medical University, Shanghai, Shanghai Municipality
  - Department of Pancreatic and Hepatobiliary Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality
  - Department of Biliary Pancreatic Surgery, Huadong Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Department of Pancreatic Surgery, Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Department of Pancreatic Surgery, Cancer Institute & Hospital, Tianjin Medical University, Tianjin, Tianjin Municipality
  - Department of General Surgery,Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang